CLINICAL TRIAL: NCT02631421
Title: Dysregulation of Lipid Metabolism and Right Ventricular Function in PAH
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Evan Brittain, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 140983
Record Dates: First submitted 2014-12-12; First posted 2015-12-16 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary Arterial Hypertension: Clinical diagnosis of pulmonary arterial hypertension
  Interventions: Procedure: Blood Sampling; Other: Cardiac MRI
- Healthy subjects and patients with other causes of PH: Patients referred for right heart catheterization who do not have PAH
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling
Other: Cardiac MRI
  Groups: Pulmonary Arterial Hypertension

SUMMARY:
Right ventricular (RV) failure is the predominant cause of death in pulmonary arterial hypertension (PAH). No RV-specific therapies are available, in part because the underlying mechanisms of RV dysfunction are poorly understood. Given the heart's preference for fatty acids (FA) as an energy source, a deeper understanding of FA metabolism may shed light on RV adaptation to elevated afterload in PAH. The purpose of this study is to test the hypothesis that defects in fatty acid metabolism are common in PAH and contribute to RV failure. The investigators will measure peripheral and transcardiac lipid and glucose metabolites in PAH patients in comparison with patients with pulmonary venous hypertension and no evidence of pulmonary hypertension. The investigators will also correlate metabolites with concurrent measurement of right ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Scheduled to undergo cardiac catheterization (right ± left heart catheterization) and/or electrophysiology study in the VHVI cardiac catheterization laboratory (CCL)/electrophysiology laboratory (EP lab)
* Hemoglobin value ≥ 10 g/dL or hematocrit of ≥ 30% (measured on clinically-indicated blood draw within 30 days or a point-of-care measurement in CCL/EP Laboratory if clinically-indicated value is not available)

Exclusion Criteria:

* Any individual that is anemic and has a hemoglobin value < 10 g/dL and hematocrit of < 30% will be excluded from the study.
* If a physician performing the procedure believes that performing the extra steps and /or acquiring the additional blood samples will delay or otherwise compromise participants' care, he/she can abandon acquisition of those data at his/her discretion.
* Contraindication to cardiac MRI (applies only to patients undergoing CMR as part of this protocol).

  * Implanted ferromagnetic material
  * Glomerular filtration rate < 60mL/min (measured on clinically-indicated blood draw within 30 days of CMR or a point-of-care measurement in the CMR Laboratory if clinically-indicated GFR is not available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAH
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Peripheral blood oleoylcarnitine in PAH versus control | At time of clinic visit, within 24 hrs prior to right heart catheritization
Percent change across the cardiac circulation of oleate and the glucose/lactate ratio. | At time of right heart catheterization
  The combination of these findings will indicate if there is a decreased reliance on FAO and and increased glycolysis

SECONDARY OUTCOMES:
Correlation of oleoylcarnitine, other acylcarnitines and free fatty acids with the homeostatic index of insulin resistance, tricuspid annular plane systolic excursion, and six minute walk distance | At time of clinic visit, within 24hrs prior to right heart catheritization
Correlation of the trans-cardiac gradient of oleate and lactate/glucose with right ventricular ejection fraction on cardiac MRI and six minute walk distance. | At time of right heart catheterization
Measurement of trans-cardiac acylcarnitines | At time of right heart catheterization
Measurement of trans-cardiac and trans-pulmonary glucose metabolites | At time of right heart catheterization
Measurement of trans-cardiac and trans-pulmonary lipid metabolites | At time of right heart catheterization
Measurement of trans-cardiac and trans-pulmonary amino acid metabolites | At time of right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, MSCI, Principal Investigator — Vanderbilt Univerisy
Locations (1):
- Vanderbilt Univeristy, Nashville, Tennessee, United States